CLINICAL TRIAL: NCT02307929
Title: Evaluation of Quality of Care - Nurse Allied Health Clinic Programme, HA
Acronym: QoC NAHC
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1189
Record Dates: First submitted 2013-08-28; First posted 2014-12-04 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Disease Management: Aging population with the need of Chronic Disease Management

SUMMARY:
In the past two decades, as a result of population aging and shifts in patient needs, we have seen an increased demand for chronic disease management (CDM) delivered in the community. The Hong Kong Government introduced six nurse allied health clinics (NAHC) programme to assist the delivery of care to facilitate the increased demand on chronic disease management (CDM) in the community, which are currently being piloted within the government funded general outpatient clinics (GOPC) of the Hospital Authority (HA). These programmes are designed to enhance CDM in primary care through patient empowerment and use of multi-disciplinary nurse and allied health led teams, and aim for secondary prevention and treat-to-target for specific health conditions. This model of care has already been established in a number of countries, namely United Kingdom, Australia, Canada and United States, where multi-disciplinary allied-health clinics, nurse practitioners and nurse-led clinics have already been integrated into routine practice in primary care (Thomas, Cullum et al. 2000; Laurant, Reeves et al. 2005).

The six NAHC programmes which have been developed to date address falls prevention (FP), continence care (CC), mental wellness (MW), wound care (WC), respiratory disease management (respiratory clinic) and medication management and compliance (MMCC). The evaluation on the QOC is an essential part of the programme in order to inform future policy. he Department of Family Medicine and Primary Care (FMPC) of the University of Hong Kong (HKU) has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the NAHC programme is achieved. Each NAHC participating clinic will be invited to complete a structured evaluation questionnaire. Anonymized data of all patients who have enrolled into the NAHC programme for more than 6 months will be included in the evaluation on the process and outcomes of care. Data on the process of care will be retrieved from the HA medical records.

In-depth study of NAHC CC programme: In order to compare the outcomes over time between subjects who have and who have not participated in the NAHC Continence Care Programme, three hundred and sixty control patients who have not been enrolled into the NAHC CC programme will be selected for the comparison in the outcomes of care. Subjects will be followed up by telephone to evaluate the effect of the programme in quality of life (QOL), patient enablement, and global rating of change in health condition at baseline , 12-month and 24-month after enrollment.

Main Outcome Measures: The primary outcomes are the proportion of participants who have received the planned process of care and have improvement in clinical outcomes.

Data Analysis: Descriptive statistics on proportions meeting the QOC criteria will be calculated. The changes in clinical, service and patient reported outcomes between baseline and discharge will assessed by paired sample t-test. The audit cycle will be repeated 4 times over a period of 5 years.

In-depth study of NAHC CC programme: the clinical outcomes between NAHC CC subjects and control group will be compared by independent sample t-test or Chi-square test.

Results: The QOC of the NAHC programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified.

Conclusion: The results of this study will provide empirical evidence on whether the HA's NAHC programmes enhance the QOC of their participating patients. This information will be used to guide service planning and policy decision making.

ELIGIBILITY:
Inclusion Criteria:

1. Falls Prevention (FP) All patients who are 60 years and above, who live in community, and who have a history of falls in the past 12 months or who are potential fallers (e.g. co-existing chronic disease, have lower limb weakness or decrease in mobility) are eligible to be recruited to the FP clinic.
2. Continence Care (CC) Patients who are >18 years old, living in the community reporting bladder or bowel problems,lower urinary tract symptoms (LUTS), constipation, and/or faecal incontinence are eligible to be recruited to the CC clinic.
3. Mental Wellness (MW) Patients who are >18 years old presenting with mild psychological health problems or who are having difficulty with coping with everyday life demands will be eligible to be recruited to the MW clinic.
4. Wound Care (WC) Patients who are >18 years old who are receiving regular wound care in the GOPC and have hard-to-heal or complicated wounds will be recruited to the WC clinic.
5. Respiratory Disease Management (respiratory clinic) Patients aged 40 years or above who are either current smokers or ex-smokers with respiratory symptoms or who are known to have Chronic obstructive pulmonary disease (COPD) are eligible to be recruited to the respiratory clinic.
6. Medication Management and Compliance Clinic (MMCC) Patients who have chronic disease with poor or questionable drug compliance, or who are on multiple medication (polypharmacy), or who are using medications or pharmaceutical devices that warrant special attention are eligible to be recruited to the MMCC programme.

Exclusion Criteria:

Continence Care (CC) Patients who live in residential care facilities will be excluded.

Mental Wellness (MW) Patients will be excluded if they live in a residential facility or have immediate psychiatric risk.

Respiratory Disease Management (respiratory clinic) Patients will be excluded if they have shortness of breath due to ischaemic heart disease or have respiratory symptoms due to infectious lung diseases.

In all programmes:

Patients will be excluded if they are unable to understand or communicate in Chinese language,or if they refuse to give consent.

In-depth study of NAHC CC programme:

NAHC participants: all new patients with LUTS. Patients will be excluded if they are unable to understand or communicate in Chinese language,or if they refuse to give consent.

Control: a modified The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form questionnaire is used to screen for patient eligibility in general-outpatient clinics. Patients will be excluded if they are aged < 18 years, could not understand Cantonese, refuse to participate, or are too ill to give consent. Patients are also excluded if they have received any service from a nurse-led primary care clinic or a specialist clinic within the past one year for his/her LUTS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in any of the programmes (fall prevention, continence care, mental wellness, wound care, respiratory disease management and medication management and compliance clinics) in Hong Kong Primary care.
Sampling Method: Probability Sample
Enrollment: 2496 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clinics that have satisfied each of the structure criteria. | Five years
  Interim analysis will evaluate the period from August, 2009 to December, 2010; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of patients who have complied with the criterion process of care. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of patients who have achieved the target of outcomes of care | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.

SECONDARY OUTCOMES:
Patient reported outcomes (PRO) measured by the change in Short Form-12v2 scores, the Patient Enablement Index and Global Rating of Change Scale scores (In-depth study of NAHC CC programme) | 2 years
  Baseline, 12-month and 24-month after the first administration of questionnaire.
Service utilization outcomes measured by GOPC consultation, Specialist Out-patient Clinics consultation, A&E and hospital attendance rates in the past 12 months.hospital attendance rates in the past 12 months. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong; W.Y. Chin, MBBS, Principal Investigator — Department of Family Medicine and Primary Care, Faculity of Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong Island, Hong Kong

REFERENCES:
- [Derived] Chin WY, Choi EP, Lam CL. The effect of timing of incentive payments on response rates for cohort study telephone interviews in primary care setting with cost-minimization analysis, a randomized controlled trial. BMC Med Res Methodol. 2015 Oct 6;15:79. doi: 10.1186/s12874-015-0073-3. PMID 26445404